CLINICAL TRIAL: NCT00802243
Title: Leflunomide Associated With Topical Corticosteroids for Bullous Pemphigoid. An Open Prospective Study
Brief Title: Leflunomide Associated With Topical Corticosteroids for Bullous Pemphigoid
Acronym: ARABUL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003545-32
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; leflunomide; corticosteroid treatment reduction; Patients are screened by: the physicians in different departments of the hospital, the liberal dermatologists and the general practicioners.; Phase I: Patients will be referred to the investigators of Dupuytren Hospital Dermatology Department.; Phase II: Patients will be referred to the investigators of Purpan (Toulouse), Haut Leveque (Pessac) and Dupuytren (Limoges) Hospitals.
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: leflunomide

SUMMARY:
Bullous pemphigoid (BP) is the most common blistering auto-immune disease of skin with an incidence estimated to 400 new cases per year. Topical corticosteroid therapy is considered the standard treatment for bullous pemphigoïd in 2002. Topical corticosteroid requires an initial large hospitalization during the acute phase and rehospitalization during relapse. The usefulness of immunosuppressive drugs have suggested by uncontrolled study.

In this way, leflunomide could be an alternative therapy, and to reduce relapse and/or resistance risks.

This study could prove the efficacity of leflunomide, associated with short time topical corticosteroids.

DETAILED DESCRIPTION:
Pre-inclusion stage: Case history, clinical examination, laboratory study, inclusion criteria checking.

Inclusion stage: Inclusion and exclusion criteria checking, clinical examination, disease follow-up, written inform consent.

Ambulatory hospitalisation, laboratory study.

Treatment and follow-up of the patients.

Clobetasol propionate cream application and leflunomide introduction.

After inclusion, the treatment will begin with 40 g topical corticosteroid per day and 20 mg leflunomide per day.

Topical corticosteroids will be progressively decreased during 5 months and stopped.

Follow-up: monthly during one year in the department of dermatology, university hospital (clinical examination, laboratory study).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 65 years old
* Bullous pemphigoid :

  * Newly diagnosed bullous pemphigoid : No treatment or topical corticosteroids therapy for less than one month
  * BP diagnosed : Resistance of the BP to the treatment or recurrence 6 months at least after diagnosis
* Follow up monthly during one year accepted
* Written Inform Consent

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Stage 1 : complete clinical remission after 6 months treatment for 9 patients at least among 15 appraisable patients.
Stage 2 : complete clinical remission after 6 months treatment for 27 patients at least among 43 appraisable patients.

SECONDARY OUTCOMES:
To determine the rate of clinical complete remission at M9 and M12.
To estimate the number of patients with immunological remission at M6, M9 and M12.
To evaluate monthly the tolerance of leflunomide.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BEDANE, MD, Principal Investigator — University Hospital, Limoges
Locations (3):
- France (3):
  - Limoges University Hospital, Limoges
  - Bordeaux University Hospital, Pessac
  - Toulouse University Hospital, Toulouse